CLINICAL TRIAL: NCT04894487
Title: The Effect of The Use of Baby Mobile Accompanied With Brhams Lullaby On The Infant's Physiologicak Parameters and Pain Level During Sternum Dressing
Brief Title: The Effects of The Use of Baby Mobile Accompanied With Brahms Lullaby On The Infants During Sternum Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Kamil KARAKAYA, Principal Investigator, RN, MSc, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15761188
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Pain, Procedural (During Sternum Dressing on Infants); Physiological Parameters During Sternum Dressing in Babies
Keywords: Sternum Dressing; Infant; Brahms Lullaby; Baby Mobile; Pain; Physiological Parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled two groups ( control group and experiment group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The babies have got sternum incision after the pediatric cardiac surgery. Experiment is about the dressing of the sternum incision. There is no extra intervention during sternum dressing at control group like routine of pediatric cardiovascular surgery intensive care clinic. Saved pain scores and physiological parameters and pain scores; just before the sternum dressing, just after sternum dressing and after the 15 minutes sternum dressing.
- THE USE OF BABY MOBILE ACCOMPANIED WITH BRAHMS LULLABIES GROUP (Experimental): Baby mobile and Brahms Lullaby started before the 10 minutes of sternum dressing process and controlled permanence of the baby mobile and Brahms Lullaby during sternum dressing. Saved pain scores and physiological parameters and pain scores; just before the sternum dressing, just after sternum dressing and after the 15 minutes sternum dressing.
  Interventions: Behavioral: THE USE OF BABY MOBILE ACCOMPANIED WITH BRAHMS LULLABY

INTERVENTIONS:
Behavioral: THE USE OF BABY MOBILE ACCOMPANIED WITH BRAHMS LULLABY — Using of baby mobile and listening Brahms Lullaby during sternum dressing process
  Arms: THE USE OF BABY MOBILE ACCOMPANIED WITH BRAHMS LULLABIES GROUP

SUMMARY:
The study was conducted experimentally in a randomized controlled manner in order to determine the effect of the use of baby mobile accompanied by Brahms Lullaby on physiological parameters and pain level during sternum dressing in babies. The research was carried out with 76 babies followed up in the Pediatric Cardiovascular Surgery Intensive Care Unit between August 2020 and February 2021 (Baby Mobile Group accompanied by Brahms Lullaby: 38, Control Group: 38). Data were collected by using the "Baby Monitoring Form" and "FLACC Pain Scale".

ELIGIBILITY:
Inclusion Criteria:

* Being 1-12 months
* Being volunteer for research
* Operated for Congenital Heart Disease
* Got Sternum incision
* No other chronic illness
* No similar surgical experiment before
* No visual impairment
* No hearing impairment
* No mental or neurological impairment
* Hospitalization experience

Exclusion Criteria:

-

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The effects of the use of baby mobile accompanied with Brahms Lullaby on the baby's pain levels during sternum dressing | 30 minutes
  FLACC Pain Scale was used for determain pain level in this research. Scale got 0 to 10 points (0 (Bad) to 10 (Good)).
The effects of the use of baby mobile accompanied with Brahms Lullaby on the baby's heart beat during sternum dressing | 30 minutes
  heart beat- bpm
The effects of the use of baby mobile accompanied with Brahms Lullaby on the baby's blood pressure sternum dressing | 30 minutes
  blood pressure- mmHg
The effects of the use of baby mobile accompanied with Brahms Lullaby on the baby's body temperature during sternum dressing | 30 minutes
  body temperature-- degrees centigrade
The effects of the use of baby mobile accompanied with Brahms Lullaby on the baby's SpO2 during sternum dressing | 30 minutes
  SpO2

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training and Research Hospital, Pediatric Cardiovascular Surgery Intensice Care Unit, Küçükçekmece, Istanbul, Turkey (Türkiye)